CLINICAL TRIAL: NCT03572452
Title: Can Sciatica Patients Due to Intervertebral Disc Herniation Avoid Surgery by Treatment Using the McKenzie Method or by Advice to Stay Active?
Brief Title: Can Sciatica Patients Avoid Surgery?
Acronym: CASPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Finland Hospital District (Other)
Collaborators: Seinajoki Central Hospital (Other); Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Sinikka Kilpikoski, PhD, PT, PhD, researcher, Central Finland Hospital District
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CentralFinlandHD
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Sciatic Nerve Compression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McKenzie - method group (Experimental): Participants will be sent to an experienced MDT therapist for therapy. They are 1) assessed clinically, 2) treated according the MDT-approach which includes home exercise program, consisting i) an educational component, and ii) an active therapy component with directional preference exercises, several times a day with sustained end range positions according to symptom response, and with avoiding aggravating positions. Participants have a maximum of 7 treatment visits. They will also have physiotherapy counselling at study entry about the good prognosis of sciatica.
  Interventions: Behavioral: McKenzie Method
- Advice to stay active group (Active Comparator): Participants enrolled into this group will receive physiotherapist's counselling at study entry for at least 60 minutes time about the good prognosis of sciatica, the spontaneous regression of the intervertebral disc herniation and pain tolerance ("natural healing"). In addition, they will get ergonomic advice and advice to stay normally active. The participants are also told to avoid bed rest and advised to continue their normal routines as actively as possible including exercise activities with limits permitted by their signs and symptoms. A two-page summary booklet related to these items will be given to them.
  Interventions: Behavioral: Advice to saty active

INTERVENTIONS:
Behavioral: McKenzie Method — Treatment according to the Mechanical Diagnosis and Therapy Approach
  Arms: McKenzie - method group
Behavioral: Advice to saty active — Physiotherapy councelling advicing to stay normally active
  Arms: Advice to stay active group

SUMMARY:
Sciatica pain is associated with a disc disorder in 85% of cases. Sciatica is shown to resolve without treatments in the majority of cases. Spontaneous regression of the intervertebral disc herniation occurs where the herniation loses its volume partly or totally without surgical interventions. It has estimated that only 5 to 20% of patients with symptomatic intervertebral disc herniation require surgery. Most trials comparing surgical trials and conservative treatments of sciatica due to intervertebral disc herniation favor surgery, because it results in earlier relief of pain. However, one year after surgery, there were only a few differences in pain and disability between surgery and conservative treatment groups. It has shown that the number of surgeries (discectomies) decreased among patients with sciatica when treated by using a mechanical diagnosis and therapy approach (MDT) also called the McKenzie method. In addition, by using the MDT method it has also been shown that sciatica patient who were clinically classified as "centralizers" had good to excellent non-surgical outcomes and many of them avoided surgery, whereas non-centralizing pain has shown to predict worse treatment outcomes, chronic low back disorder and disability. Further, patients who do not have centralization will be 6 times more likely to undergo surgery.The primary aim of this multicenter randomized clinical trial is to find out how many patients with sciatica due to intervertebral disc herniation with radicular symptoms for at least 6 weeks, and who are on the waiting list for surgery, avoid surgery by treatment using the McKenzie method compared to advice to stay active. Secondary aims are to compare the patients' self-reported outcomes such as low back and leg pain intensity, disability, work ability, sick-leave days, fear avoidance beliefs, kinesiophobia, depression and quality of life. The outcomes are measured at baseline, two and three months in the non-surgical patients. In addition, in the patients who have surgery the outcomes are measured at baseline and the day before and one month after surgery. Follow-up measurements are at 12 and 24 months

DETAILED DESCRIPTION:
One hundred seventy two (N=172) patients with sciatica for at least six weeks with radicular pain below the knee will be involved this study. The patients with non-urgent referrals due to sciatica symptoms will be directed to specialized medical care hospitals (the district central hospitals of Central Finland and South Ostrobothnia and the University hospital of Kuopio, Finland) to the physiatrists and orthopedic outpatient clinics for further investigations for possible surgery. The patient will be seen for a doctor's examination within a week. If the clinical examination reveals that a patient needs spinal disc herniation surgery, and the patient is willing to undergo surgery, they will be referred for X-ray imaging if it has not already been done in basic health care, in accordance with the regular treatment procedure, and to an MRI scan.

While patients are waiting for their MRI scan, they will undergo a clinical McKenzie-based mechanical assessment and be put into sub-groups of "centralizers"or "non-centralizers". These will be randomly assigned into a McKenzie group and into an advice to stay active group. Based on their MRI findings and clinical signs and symptoms they will be assigned to surgery or continue their non-surgical treatments. If the MRI scan does not reveal a spinal disc herniation finding that fulfills the criteria of the study, the patient is removed from the study in accordance with the selection criteria, regardless of whether they belong to the MDT or advice to stay active group, and their treatment will continue according to the hospital's normal procedures.

ELIGIBILITY:
Inclusion Criteria: The participants are 18 - 60-year-old Finnish speaking sciatica patients for whom magnetic resonance imaging confirmed disc herniation compressing a nerve root canal, and who have related symptoms radiating to the lower limb +/- neurological disorders. Their sciatica has lasted at least 6 weeks.

Exclusion Criteria:

Pregnancy, previous surgery or treated by using MDT- method, fibromyalgia, signs of serious diseases or "red-flags" symptoms. Symptoms indicating the Cauda Equina Syndrome (CES) or lower limb palsy that hinders normal functioning, previous injury from a car accident or a high fall, or osteoporotic fractures for the elderly, cancer anamnesis, tumor, or inflammation, general symptoms such as fever, chills, or losing weight for an unknown reason, back problems complicated by other serious diseases such as polyneuropathy, neurological diseases, circulatory brain diseases, central spinal stenosis, myelopathy, syringomyelia, and long-term neuropathic pain not related to sciatica, unwillingness to undergo surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients who avoided surgery | Changes are reported from baseline to short term (3 months), longer term (12months) and in long term (24months) follow-ups
  Number of patients who avoided surgery treated by using the McKenzie- method or by advice to stay active

SECONDARY OUTCOMES:
Pain Intensity | Changes are reported from baseline to short term (3 months), longer term (12months) and in long term (24months) follow-ups
  Low back and leg pain intensity reported with Visual Analog Scale (VAS) (0 - 100mm scales, 0 mm = no pain, 100mm = worst possible pain).
Disability | Changes are reported from baseline to short term (3 months), longer term (12months) and in long term (24months) follow-ups.
  Disability is reported with Oswestry disability index Finnish version 2.0 total score (scale 0-100%): 0= minimal disability, 100 = bed-bound or exaggeration of symptoms.
Health-Related Quality of Life | Changes are reported from baseline to longer term (12months) and in long term (24months) follow-ups
  Quality of life is assessed with the SF-36.These eight scale scores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores equals more disability, higher scores equals less disability. Physical and mental components will be calculated separately.

OTHER OUTCOMES:
Fear Avoidance | Changes are reported from baseline to short term (3 months), longer term (12months) and in long term (24months) follow-ups
  Fear-avoidance beliefs about physical activity and work was measures with the Fear Avoidance Beliefs Questionnaire (FABQ). It consists of 16 questions, for each statement has a 7-point Likert scale with scoring alternatives ranging from "0 = completely disagree" to "6 = completely agree".
Kinesiophobia | Changes are reported from baseline to short term (3 months), longer term (12months) and in long term (24months) follow-ups.
  The fear to move was assessed with the Tampa Scale for Kinesiophopia (TSK) questionnaire. It comprises 17 items assessing the subjective rating of kinesiophopia. Each item has a 4-point Likert scale with scoring alternatives ranging from "strongly disagree" to "strongly agree".
Depression | Changes are reported from baseline to short term (3 months), longer term (12months) and in long term (24months) follow-ups.
  Depression during last month is measured with the Depression Scale (DEPS) questionnaire.This self-rating depression scale in Finnish consists of 10 items. Each item has a 4-point scale with alternatives ranging from "0 = not at all" to "3 = very much".
Work ability | Changes are reported from baseline to short term (3 months), longer term (12months) and in long term (24months) follow-ups.
  Work ability is measured with the Visual Analogue Scale (VAS) from 0 to 100mm scales (0 mm = completely able to work and 100mm = unable to work).
Sick leave | Changes are reported from baseline to short term (3 months), longer term (12months) and in long term (24months) follow-ups.
  Number of sick leave days

CONTACTS AND LOCATIONS:
Overall Officials: Jari Ylinen, MD,PhD., Study Director — Central Finland HD
Locations (1):
- Central Finland Central Hospital,, Jyväskylä, Central Finland, Finland

IPD SHARING:
Plan to Share IPD: No